CLINICAL TRIAL: NCT07230119
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase 3 Study to Evaluate the Efficacy and Safety of Zovaglutide in Adults With Overweight or Obesity.
Brief Title: A Study of Zovaglutide in Subjects With Overweight or Obesity (HORIZON-1)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BJQL-ZT002-3001
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Overweight , Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zovaglutide dose 1 (Experimental): administered subcutaneously (SC), Q4W
  Interventions: Drug: Zovaglutide dose 1
- Zovaglutide dose 2 (Experimental): administered subcutaneously (SC), Q4W
  Interventions: Drug: Zovaglutide dose 2
- Placebo (Placebo Comparator): Administered subcutaneously (SC), Q4W
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zovaglutide dose 1 — administered subcutaneously (SC), Q4W
  Other Names: ZT002 Injection
  Arms: Zovaglutide dose 1
Drug: Zovaglutide dose 2 — administered subcutaneously (SC), Q4W
  Other Names: ZT002 Injection
  Arms: Zovaglutide dose 2
Drug: Placebo — administered subcutaneously (SC), Q4W
  Arms: Placebo

SUMMARY:
This study will evaluate the percentage change in body weight from baseline and proportion of subjects achieving ≥ 5% weight loss from baseline after 52 weeks of treatment with Zovaglutide in subjects with overweight/obesity.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female subjects aged≥18years and≤75 years at the time of signing the ICF.
* 2.At screening and prior to randomization, BMI must meet one of the following criteria:

  1. BMI≥28kg/m²regardless of comorbidities；
  2. BM≤24 kg/m² and<28 kg/m², with at least one of the following comorbidities: prediabetes, hypertension, dyslipidemia, fatty liver disease, obstructive sleep apnea syndrome due to overweight, or weight-bearing joint pain.
* 3.Weight change due to diet and exercise alone within 3 months prior to screening and randomization did not exceed 5%.

Exclusion Criteria:

* 1.Previously diagnosed obesity caused by monogenic mutations, other diseases, or medications.
* 2.Previous diagnosis of diabetes; or HbA1c ≥ 6.5% or fasting blood glucose ≥ 7.0 mmol/L at screening.
* 3.Used of medicines or treatments that affect weight within 3 months prior to screening.
* 4.History of acute or chronic pancreatitis, or pancreatic injury.
* 5.History of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine neoplasia (MEN2) in personal or family history.
* 6.History of depression/anxiety disorder, or prior diagnosis of moderate-to-severe anxiety/depressive state, or history of severe psychiatric disorders;
* 7. PHQ-9 scale score is ≥ 15 at screening;
* 8. Screening C-SSRS questionnaire suicide ideation response of "Category 4 or 5," or any "yes" response to suicidal behavior questions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Estimated)
Dates: Start 2026-03-08 (Estimated); Primary Completion 2027-05-29 (Estimated); Study Completion 2027-06-26 (Estimated)

PRIMARY OUTCOMES:
Change in body weight(%) | baseline (week 0) to week 52
Proportion of subjects achieving ≥ 5% weight loss | 52 weeks

SECONDARY OUTCOMES:
Proportion of subjects achieving ≥10% weight loss | week 52
Proportion of subjects achieving ≥15% weight loss. | week 52
Proportion of subjects achieving ≥20% weight loss. | week 52
Change in body weight (kg) | Baseline (week 0) to week 52
Change in BMI (kg/m²) | Baseline (week 0) to week 52
Change in waist circumference (cm) | Baseline (week 0) to week 52
Change in hip circumference (cm) | Baseline (week 0) to week 52
Number of Treatment Emergent Adverse Events (TEAEs) | Baseline (week 0) to week 56
Number of Serious Adverse Events (SAEs) | Baseline (week 0) to week 56
Positive rate of anti-drug antibodies (ADA). | Baseline (week 0) to week 56
Positive rate of neutralizing antibodies (Nab) | Baseline (week 0) to week 56

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD, Principal Investigator — Peking University People's Hospital
Locations (25):
- China (25):
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Guangzhou Red Cross Hospital, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - The Second Affiliated Hospotal of Guangxi Medical University, Nanning, Guangxi
  - Handan First Hospital, Handan, Hebei
  - Hebei Petro China Cental Hospital, Langfang, Hebei
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Second Hospital of Hebei Medical University, Shijiangzhuang, Hebei
  - The Fourth Affiliated Hospital Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Luoyang Third People's Hospital, Luoyang, Henan
  - The First Affiliated of Nanyang Medical College, Nanyang, Henan
  - Nanyang Second People's Hospital, Nanyang, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - Yueyang People's Hospital, Yueyang, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Xi'an Daxing Hospital, Xi’an, Shanxi
  - Peking University People's Hospital, Beijing